CLINICAL TRIAL: NCT00292864
Title: Phase 1 Open-Label, Multicenter, Dose-Escalation Clinical Study of the Safety and Tolerability of SNS-032, a Novel Cyclin-Dependent Kinase Inhibitor, Administered to Patients With Select Advanced Solid Tumors
Brief Title: Safety Assessment of One-hour Infusions of SNS-032 for the Treatment of Select Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0007
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Tumors
Keywords: Cancer; Carcinoma; Adenocarcinoma; Tumor; Advanced solid tumors
MeSH Terms: conditions — Neoplasms; Carcinoma; Adenocarcinoma | interventions — N-(5-(((5-(1,1-dimethylethyl)-2-oxazolyl)methyl)thio)-2-thiazolyl)-4-piperidinecarboxamide

INTERVENTIONS:
Drug: SNS-032 Injection

SUMMARY:
The purpose of this study is to assess the safety and tolerability of one-hour infusions given once daily for 5 consecutive days in a 21-day treatment cycle; to define a recommended phase 2 dose; and to learn more about the clinical activity of SNS-032.

DETAILED DESCRIPTION:
Other objectives of this study include measuring pharmacokinetics (how long the drug can be measured in the body), preliminary evaluation of biomarkers to see how the levels of certain proteins change after administration of SNS-032; assessment of the effects of SNS-032 on QT interval.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Advanced, progressing solid tumor that has no cure

  * In Stage 1, any advanced solid malignancy
  * In Stage 2, advanced breast cancer, melanoma, or non-small cell lung cancer (NSCLC)
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Recovered from radiation therapy that may have been given in the last 21 days
* Recovered from surgery

Exclusion Criteria:

* Prior exposure to SNS-032 (previously known as BMS-387032)
* Pregnant or breastfeeding
* Women or male partners of women who are able to have children but are unwilling to use an approved, effective means of birth control
* Took part in another clinical trial during the last 21 days
* Abnormal lab values for serum potassium, hemoglobin, neutrophils, platelets, creatinine, AST, ALT, or total bilirubin
* Brain metastases, if patient is not neurologically stable or has needed corticosteroids or anticonvulsants at anytime within the 28 day period before enrollment.
* Other active malignancies
* Prior pelvic radiation therapy to ≥ 25% of bone marrow reserve
* Any other condition that would keep the patient from safely taking part in the clinical trial

Please note: There are additional inclusion/exclusion criteria for this study. Please contact the study center for additional information and to determine if all study criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-01; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety
Tolerability

SECONDARY OUTCOMES:
Pharmacokinetic profile
Effect on QT interval
Potential biomarkers
Anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Adelman, MD, Study Director — Sunesis Pharmaceuticals
Locations (6):
- United States (6):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - University of California Davis Medical Center, Davis, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148